CLINICAL TRIAL: NCT01024023
Title: Hull - Early Walking Aids for Transtibial Amputees - Does an Articulated Knee Have Benefits? A Randomised Controlled Trial
Brief Title: Hull Early Walking Aids for Transtibial Amputees - Randomised Control Trial (HEART)
Acronym: HEART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Hull (Other)
Collaborators: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Amanda Hancock / Physiotherapy Clinical Manager Inpatients CHH, Physiotherapy Department, Castle Hill Hospital, Hull & East Yorkshire Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R0081
Record Dates: First submitted 2009-11-25; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Unilateral Trans-tibial Amputees
Keywords: Early Walking Aid; Amputee; Trans-tibial; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PPAM Aid (Active Comparator): Suitable participants randomised to the treatment arm will receive the non articulated pneumatic early walking aid and rehabilitation physiotherapy will be commenced immediately. Physiotherapy will continue after they receive their definitive prosthesis till they are comfortable and safe using it, at which stage they will be discharged and no further follow up will be performed.
  Interventions: Device: EWA
- AMA Aid (Active Comparator): Suitable participants randomised to the treatment arm will receive the articulated early walking aid and rehabilitation physiotherapy will be commenced immediately. Physiotherapy will continue after they receive their definitive prosthesis till they are comfortable and safe using it, at which stage they will be discharged and no further follow up will be performed.
  Interventions: Device: EWA

INTERVENTIONS:
Device: EWA — Suitable participants randomised to the treatment arm to receive early walking aid and rehabilitation physiotherapy will be commenced immediately. Physiotherapy will continue after they receive their definitive prosthesis till they are comfortable and safe using it, at which stage they will be discharged and no further follow up will be performed.
  Other Names: Pneumatic Post Amputation Mobility Aid - Ortho Europe Ltd,UK; Amputee Mobility Aid - Ortho Europe Ltd,UK

SUMMARY:
Early walking aids are routinely used in UK for rehabilitation of patients with below knee amputations. The two main walking aids used commonly in practice include the non-articulated Pneumatic Post Amputation Mobility Aid (PPAM)and the Articulated Amputee Mobility Aid (AMA). There is no published evidence on whether the articulated walking aid improves knee control and shortens delivery time. This study was designed to test the hypothesis that an articulated early walking aid has benefit to transtibial amputee compared to non-articulated early walking aid.

DETAILED DESCRIPTION:
Physiotherapists in the UK routinely use Early Walking Aids (EWA's) to enable the lower limb amputee to start to walk again as early as 5 days post amputation (Lein S. 1992). An EWA has many benefits including a reduction in oedema (Reith et al, 1992) early gait and balance training in preparation for using a prosthesis. The two EWA's most commonly used in the UK for transtibial amputees are the Pneumatic Post Amputation Mobility aid (PPAM) and the Amputee Mobility Aid (AMA). A comparison of the PPAM aid and the AMA undertaken by Longmore T (1997) reported no significant difference in energy cost, comfort or ease of use. Scott et al (2000) found the AMA to have higher interface pressures than the PPAM aid. There is however no known published evidence on whether an articulated EWA improves active knee control following prosthetic delivery and therefore shortens rehabilitation time. In addition there is no known published evidence of the effect on quality of life with the two different EWA's.

Hypothesis: An articulated Early walking aid has benefit to the transtibial amputee compared to a non- articulated EWA.

The purpose of this proposed research is to investigate whether there are any benefits to patients in using an articulated EWA.

The study will use EMG and gait analysis to determine the potential of each of the two EWA's to re-educate gait in a way that is comparable with the gait exhibited when the subject subsequently begins to use a prosthesis thus shortening rehabilitation time. Quality of life indicators will be used to determine the impact on the patient and, in addition, the length of time taken to full rehabilitation will be considered.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the trial if they:

* Have had a unilateral transtibial amputation but not yet received a prosthesis
* Are expected to receive a functional prosthesis
* Are at least 18 years of age
* Are able to tolerate and use an early walking aid
* Are able to be able to walk a distance of 4 metres
* Will attend Hull and East Yorkshire Hospitals NHS Trust for prosthetic rehabilitation.
* Meet the manufacturers recommendations for using the EWA's

Exclusion Criteria:

Patients will be excluded from the trial if they:

* Have had a major amputation of the contra lateral limb.
* Are not expected to receive a functional prosthesis
* Were unable to walk, prior to their amputation, due to a medical condition e.g. spinal injury, stroke or rheumatoid arthritis
* Are unable to follow instructions and/or participate in a programme of rehabilitation.
* Do not consent to participate in the study.
* Do not meet the manufacturers recommendations for using the EWA's

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-12; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Kinetic and kinematic comparison of the influence of 2 different EWAs on the transfer to prosthetic rehabilitation. | Outcomes will be measured at baseline, time of EWA fitting, prosthesis fitting, 2 week post prosthesis fitting &on discharge from physiotherapy ensuring safe prosthesis use. Final visit will vary with each patient and will be analysed with outcomes.

SECONDARY OUTCOMES:
Quality of life measurements | Outcomes will be measured at baseline, time of EWA fitting, prosthesis fitting, 2 week post prosthesis fitting &on discharge from physiotherapy ensuring safe prosthesis use. Final visit will vary with each patient and will be analysed with outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Hancock, MSc, Principal Investigator — Department of Physiotherapy, Hull & East Yorkshire Hospitals NHS Trust; Ian C Chetter, MB ChB, FRCS, Study Director — University of Hull
Locations (3):
- United Kingdom (3):
  - Academic Vascular Surgical Unit, University of Hull, Hull, Humberside
  - Physiotherapy Department, Hull & East Yorkshire Hospitals NHS Trust, Hull, Humberside
  - Department of Sports, Health & Exercise Science, University of Hull, Hull, Humberside

REFERENCES:
- [Background] Barnett C, Vanicek N, Polman R, Hancock A, Brown B, Smith L, Chetter I. Kinematic gait adaptations in unilateral transtibial amputees during rehabilitation. Prosthet Orthot Int. 2009 Jun;33(2):135-47. doi: 10.1080/03093640902751762. PMID 19367517